CLINICAL TRIAL: NCT02199145
Title: Indication and Response to Immunosuppressive Treatment in Membranous Nephropathy : Role of Anti-mouse PLA2R1 ELISA
Brief Title: Role of Anti-mouse PLA2R1 ELISA in Membranous Nephropathy
Acronym: SOURIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-AOI-05
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood and urine analysis (Other): creatinine, albumin, blood electrolytes, proteinuria /creatinine in sample 1 assay Ac anti-PLA2R1 on 3 ELISA (human, rabbit and mouse)
  Interventions: Procedure: Blood and urine analysis

INTERVENTIONS:
Procedure: Blood and urine analysis — creatinine, albumin, blood electrolytes, proteinuria / creatinine in sample 1 assay Ac anti-PLA2R1 on 3 ELISA (human, rabbit and mouse)

SUMMARY:
Membranous Nephropathy (MN) is an auto-immune kidney disease and a common cause of nephrotic syndrome. About 30% of MN patients progress to end-stage kidney disease (ESKD) while 30% undergo spontaneous remission. The phospholipase A2 receptor (PLA2R1) is the major auto-antigen in idiopathic MN. Anti-PLA2R1 autoantibodies are found during the active phase of MN. Predictors of disease progression include high titers of anti-PLA2R1 autoantibodies and serum creatinine levels at presentation, as well as decline in renal function during the first six months of follow-up. Investigators identified new prognostic factors in a cohort of 41 idiopathic MN patients with nephrotic syndrome and anti-PLA2R1 autoantibodies at the time of presentation. During a follow-up of at least 36 months, 21 patients had a persistent nephrotic syndrome (group A) and 20 showed partial or total remission (group R). We first measured the cross-reactivity of their sera at the time of presentation to human, rabbit and mouse recombinant PLA2R1 by western blot. All patients exhibited reactivity against human and rabbit PLA2R1, but only some of them did against mouse PLA2R1. These results suggest the presence of distinct epitopes that are differentially conserved among PLA2R1 orthologs.Investigators then set-up three parallel ELISAs using human, rabbit and mouse recombinant PLA2R1. All 41 MN patients showed activity in human and rabbit ELISAs at presentation but only 32 of them (78%) in mouse ELISA.They finally analyzed the association between anti-PLA2R1 titers at presentation in the different ELISAs and the subsequent clinical outcome. The mean anti-PLA2R1 activity was significantly different between group A and R in mouse ELISA but not in human and rabbit ELISA. Patients with anti-mouse PLA2R1 activity over 605 RU (relative unit)/ml showed a significantly lower survival without doubling of serum creatinine or ESKD , but patients in the highest tertile of anti-PLA2R1 activity in rabbit and human ELISA did not show a significant increased risk of renal failure progression. The results suggest that the specific detection of particular anti-PLA2R1 autoantibodies using the novel anti-mouse PLA2R1 ELISA can identify MN patients at risk for ESKD. The aim is to confirm these result on a prospective cohort.

DETAILED DESCRIPTION:
Membranous Nephropathy (MN) is an auto-immune kidney disease and a common cause of nephrotic syndrome. About 30% of MN patients progress to end-stage kidney disease (ESKD) while 30% undergo spontaneous remission. The phospholipase A2 receptor (PLA2R1) is the major auto-antigen in idiopathic MN. Anti-PLA2R1 autoantibodies are found during the active phase of MN [2,3]. Predictors of disease progression include high titers of anti-PLA2R1 autoantibodies and serum creatinine levels at presentation, as well as decline in renal function during the first six months of follow-up. Investigators identified new prognostic factors in a cohort of 41 idiopathic MN patients with nephrotic syndrome and anti-PLA2R1 autoantibodies at the time of presentation. During a follow-up of at least 36 months, 21 patients had a persistent nephrotic syndrome (group A) and 20 showed partial or total remission (group R). We first measured the cross-reactivity of their sera at the time of presentation to human, rabbit and mouse recombinant PLA2R1 by western blot. All patients exhibited reactivity against human and rabbit PLA2R1, but only some of them did against mouse PLA2R1. These results suggest the presence of distinct epitopes that are differentially conserved among PLA2R1 orthologs. We then set-up three parallel ELISAs using human, rabbit and mouse recombinant PLA2R1. All 41 MN patients showed activity in human and rabbit ELISAs at presentation but only 32 of them (78%) in mouse ELISA.

Investigators finally analyzed the association between anti-PLA2R1 titers at presentation in the different ELISAs and the subsequent clinical outcome. The mean anti-PLA2R1 activity was significantly different between group A and R in mouse ELISA in both univariate and multivariate analyses (p =0.006 and p =0.02, respectively) but not in human and rabbit ELISAs. An analysis of the mouse ELISA titers defines a threshold of 605 RU/ml above which 100% of patients had a poor prognosis, but no such threshold could be defined in rabbit and human ELISA. Patients with anti-mouse PLA2R1 activity over 605 RU/ml showed a significantly lower survival without doubling of serum creatinine or ESKD (p=0.002 using the log-rank test), but patients in the highest tertile of anti-PLA2R1 activity in rabbit and human ELISAs did not show a significant increased risk of renal failure progression. The results suggest that the specific detection of particular anti-PLA2R1 autoantibodies using the novel anti-mouse PLA2R1 ELISA can identify MN patients at risk for ESKD. The aim is to confirm these result on a prospective cohort.We propose to measure on a prospective cohort at the time of MN diagnosis if high titer of anti-mPLA2R1 Ab (anti-mouse phospholipase A2 receptor1 antibodies) is associated with nephrotic proteinuria (over 3.5 g/g) or increased of creatininemia over 30% at month 6, 12 and 18. An ancillary study will try to characterised the nephrogenic epitope conserved between human, rabbit and mouse.

Each patient with nephrotic syndrome should benefit of a kidney biopsy. For each patient we will conserved 2 dry tubes frozen at the time of biopsy. If we confirm the diagnosis of MN with anti-PLA2R1 Ab, we propose to the patient to be included in this study. He will have a visit every months for the first three months and every three months after, with collection of the following: blood pressure, weight, creatinine, albumin, blood electrolytes, proteinuria / creatinine in sample 1 assay Ac anti-PLA2R1 on 3 ELISA (human, rabbit and mouse) In case of persistent refractory nephrotic syndrome after 6 months, or the appearance of a 30% increase in serum creatinine, treatment with rituximab (2 × 1 g IV 15 days) will be proposed. Clinical and biological monitoring will be continued every 3 months for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients with MN stade I-II confirmed by kidney biopsy
* Patients with MDRD>30 ml/mn/1.73m2
* Patients with anti-PLA2R1 antibodies
* Effective Contraception for women of childbearing age

Exclusion Criteria:

* Patients minors
* Patients refusing to participate in the study
* Patients with secondary MN (systemic Lupus, hepatitis B virus, hepatitis C virus or cancer)
* Pregnant women: a urine pregnancy test will be performed for women of childbearing age. The results will be communicated to the patient by a doctor of his choice.
* Persons deprived of liberty (administrative or judicial)
* Persons under guardianship
* People may not understand the research
* Persons under guardianship, under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline Creatininemia level | at 6, 12 and 18 months
  30% increase in creatininemia after 6 months of symptomatic treatment with RAAS blocker

SECONDARY OUTCOMES:
Remission rate in MN | at 12 months
  Remission rate in MN one year after Rituximab with absence of nephrotic syndrome and renal insufficiency (estimated by MDRD> 60 ml/min/1, 73m2).
  (MDRD=Modification of the Diet in Renal Disease)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara SEITZ-POLSKI, PhD, Principal Investigator — Nice University Hospital
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - AP-HM, Marseille
  - Nephrology Department, Nice University Hospital, Nice

REFERENCES:
- [Derived] Teisseyre M, Cremoni M, Boyer-Suavet S, Crepin T, Benzaken S, Zorzi K, Esnault V, Brglez V, Seitz-Polski B. Rituximab Immunomonitoring Predicts Remission in Membranous Nephropathy. Front Immunol. 2021 Oct 13;12:738788. doi: 10.3389/fimmu.2021.738788. eCollection 2021. PMID 34721403
- [Derived] Seitz-Polski B, Dahan K, Debiec H, Rousseau A, Andreani M, Zaghrini C, Ticchioni M, Rosenthal A, Benzaken S, Bernard G, Lambeau G, Ronco P, Esnault VLM. High-Dose Rituximab and Early Remission in PLA2R1-Related Membranous Nephropathy. Clin J Am Soc Nephrol. 2019 Aug 7;14(8):1173-1182. doi: 10.2215/CJN.11791018. Epub 2019 Jul 24. PMID 31340979